CLINICAL TRIAL: NCT05423964
Title: Impact of Artificial Intelligence on Trainee Adenoma Detection Rate
Brief Title: Impact of AI on Trainee ADR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, James Buxbaum, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-21-00094
Record Dates: First submitted 2022-04-26; First posted 2022-06-21 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Adenoma; Adenoma Colon; Colorectal Cancer
MeSH Terms: conditions — Adenoma; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial Intelligence Endoscopy Room (Active Comparator): The fellows will be randomized on a daily basis to perform colonoscopies in a room with AI (intervention)
  Interventions: Diagnostic Test: AI use in Endoscopy Room
- Non-Artificial Intelligence Endoscopy Room (Active Comparator): The fellows will be randomized on a daily basis to perform colonoscopies in a non-AI endoscopy room (standard of care).
  Interventions: Other: Non-AI use Standard of Care endoscopy room

INTERVENTIONS:
Diagnostic Test: AI use in Endoscopy Room — The use of AI versus no AI in comparing the detection of adenomas during Endoscopy procedures.
  Arms: Artificial Intelligence Endoscopy Room
Other: Non-AI use Standard of Care endoscopy room — Non-AI use in comparing the detection of adenomas during Endoscopy procedures.
  Arms: Non-Artificial Intelligence Endoscopy Room

SUMMARY:
Adenoma detection rate (ADR) is a validated quality metric for colonoscopy with higher ADR correlated with improved colorectal cancer outcomes. Artificial intelligence (AI) can automatically detect polyps on the video monitor which may allow endoscopists in training to improve their ADR. Objective and Purpose of the study: Measure the effect of AI in a prospective, randomized manner to determine its impact on ADR of Gastroenterology trainees.

DETAILED DESCRIPTION:
Our objective is to determine the impact of AI on the adenoma detection rate of Gastroenterology trainees. The secondary aim of this quality improvement study is to determine the impact of AI based endoscopy on the rate of recording of quality improvement metrics versus historical performance in our program.

Fellows will undergo educational session prior to the start of study, describing commonly used metrics for assessing quality of colonoscopy and how to use the artificial intelligence software. Gastroenterology fellows will be consented for the study prior to initiation. The fellows will be randomized on a daily basis to perform colonoscopies in a room. Outcomes will measure the effects of AI in fellows

ELIGIBILITY:
Inclusion Criteria:

* All Gastroenterology fellows at USC performing Endoscopies will be included in the study.

Exclusion Criteria:

* If fellows refuse informed consent they will be excluded.
* Procedures performed in the intensive care unit or the operating room will not be counted toward the study metrics as the AI system will only be available in the endoscopy unit.
* If procedures are performed only by faculty, in which the fellow is not the primary operator, they will not be used for study metrics.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Average adenoma detection rate | Throughout study, an average of 2 years
  Adenoma detection rate with and without AI

SECONDARY OUTCOMES:
Average of polyps detection rate | Through out study, an average of 2 years
  Polyp detection rate with and without AI

CONTACTS AND LOCATIONS:
Overall Officials: James L Buxbaum, MD, Principal Investigator — University of Southern California
Locations (1):
- LAC+USC Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Fedewa SA, Ahnen DJ, Meester RGS, Barzi A, Jemal A. Colorectal cancer statistics, 2017. CA Cancer J Clin. 2017 May 6;67(3):177-193. doi: 10.3322/caac.21395. Epub 2017 Mar 1. PMID 28248415
- [Background] Winawer SJ, Zauber AG, Ho MN, O'Brien MJ, Gottlieb LS, Sternberg SS, Waye JD, Schapiro M, Bond JH, Panish JF, et al. Prevention of colorectal cancer by colonoscopic polypectomy. The National Polyp Study Workgroup. N Engl J Med. 1993 Dec 30;329(27):1977-81. doi: 10.1056/NEJM199312303292701. PMID 8247072
- [Background] Zauber AG, Winawer SJ, O'Brien MJ, Lansdorp-Vogelaar I, van Ballegooijen M, Hankey BF, Shi W, Bond JH, Schapiro M, Panish JF, Stewart ET, Waye JD. Colonoscopic polypectomy and long-term prevention of colorectal-cancer deaths. N Engl J Med. 2012 Feb 23;366(8):687-96. doi: 10.1056/NEJMoa1100370. PMID 22356322
- [Background] Rex DK, Boland CR, Dominitz JA, Giardiello FM, Johnson DA, Kaltenbach T, Levin TR, Lieberman D, Robertson DJ. Colorectal Cancer Screening: Recommendations for Physicians and Patients from the U.S. Multi-Society Task Force on Colorectal Cancer. Am J Gastroenterol. 2017 Jul;112(7):1016-1030. doi: 10.1038/ajg.2017.174. Epub 2017 Jun 6. PMID 28555630
- [Background] Corley DA, Jensen CD, Marks AR, Zhao WK, Lee JK, Doubeni CA, Zauber AG, de Boer J, Fireman BH, Schottinger JE, Quinn VP, Ghai NR, Levin TR, Quesenberry CP. Adenoma detection rate and risk of colorectal cancer and death. N Engl J Med. 2014 Apr 3;370(14):1298-306. doi: 10.1056/NEJMoa1309086. PMID 24693890
- [Background] Abadir AP, Ali MF, Karnes W, Samarasena JB. Artificial Intelligence in Gastrointestinal Endoscopy. Clin Endosc. 2020 Mar;53(2):132-141. doi: 10.5946/ce.2020.038. Epub 2020 Mar 30. PMID 32252506
- [Background] Urban G, Tripathi P, Alkayali T, Mittal M, Jalali F, Karnes W, Baldi P. Deep Learning Localizes and Identifies Polyps in Real Time With 96% Accuracy in Screening Colonoscopy. Gastroenterology. 2018 Oct;155(4):1069-1078.e8. doi: 10.1053/j.gastro.2018.06.037. Epub 2018 Jun 18. PMID 29928897
- [Background] Repici A, Badalamenti M, Maselli R, Correale L, Radaelli F, Rondonotti E, Ferrara E, Spadaccini M, Alkandari A, Fugazza A, Anderloni A, Galtieri PA, Pellegatta G, Carrara S, Di Leo M, Craviotto V, Lamonaca L, Lorenzetti R, Andrealli A, Antonelli G, Wallace M, Sharma P, Rosch T, Hassan C. Efficacy of Real-Time Computer-Aided Detection of Colorectal Neoplasia in a Randomized Trial. Gastroenterology. 2020 Aug;159(2):512-520.e7. doi: 10.1053/j.gastro.2020.04.062. Epub 2020 May 1. PMID 32371116
- [Background] Calderwood AH, Jacobson BC. Comprehensive validation of the Boston Bowel Preparation Scale. Gastrointest Endosc. 2010 Oct;72(4):686-92. doi: 10.1016/j.gie.2010.06.068. PMID 20883845
- [Background] Kaminski MF, Regula J, Kraszewska E, Polkowski M, Wojciechowska U, Didkowska J, Zwierko M, Rupinski M, Nowacki MP, Butruk E. Quality indicators for colonoscopy and the risk of interval cancer. N Engl J Med. 2010 May 13;362(19):1795-803. doi: 10.1056/NEJMoa0907667. PMID 20463339
- [Background] Jovani M, Campbell EJ, Hur C, Joshi AD, Nishioka NS. Effect of video monitor size on polyp detection: a prospective, randomized, controlled trial. Gastrointest Endosc. 2019 Aug;90(2):254-258.e2. doi: 10.1016/j.gie.2019.03.1172. Epub 2019 Apr 12. PMID 30986402
- [Derived] Chang PW, Nguyen DD, Kong N, Wang D, Wang S, Ong J, Amini MM, Sharma N, Bui A, Bakr O, Bruce D, Lee H, Dodge JL, Sahakian AB, Buxbaum JL. Impact of artificial intelligence-assisted colonoscopy on gastroenterology fellow performance: a pragmatic randomized controlled trial. Gastrointest Endosc. 2025 Sep 27:S0016-5107(25)02063-2. doi: 10.1016/j.gie.2025.09.045. Online ahead of print. PMID 41022225